CLINICAL TRIAL: NCT00237393
Title: A Randomized, Placebo-Controlled Trial of Quetiapine (Seroquel) Monotherapy in the Treatment of PTSD
Brief Title: Quetiapine Treatment for Post-Traumatic Stress Disorder (PTSD)
Acronym: PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Collaborators: AstraZeneca (Industry)
Responsible Party: Mark B. Hamner, MD, Ralph H. Johnson VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0058; HR-10762
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2005-10

CONDITIONS: PTSD
Keywords: PTSD; Posttraumatic stress disorder; Treatment; Quetiapine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Quetiapine
  Interventions: Drug: Quetiapine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine — Dosage initiated at 25 mg HS with gradual titration to target dose of 400 mg HS, up to maximum of 800 mg HS.
  Arms: 1
Drug: Placebo — Dosage initiated at 25 mg HS with gradual titration to target dose of 400 mg HS, up to maximum of 800 mg HS.
  Arms: 2

SUMMARY:
The purpose of the study is to determine if quetiapine is effective in the treatment of PTSD.

DETAILED DESCRIPTION:
Objective: To assess the impact of quetiapine on core PTSD symptoms and associated psychiatric comorbidity including depressive and positive and negative psychotic symptoms.

Research Design: 12-week, double-blind, placebo-controlled, randomized, fixed-flexible dose trial of quetiapine monotherapy.

Intervention: Eligible patients will be randomized to receive quetiapine starting at 25 mg daily or matching placebo. Dose adjustments (to a minimum of 50 mg or a maximum of 800 mg), will be made at the investigator's discretion and according to patient's clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older of any ethnic background meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for PTSD.
* Score of at least 50 on the CAPS-SX at baseline.
* Competent to give informed consent.
* If female, patient should be using a medically approved contraceptive, or not otherwise be of childbearing potential.
* Patients who have not taken medications or herbal remedies for a psychiatric indication within one week prior to the randomized phase.
* Other medications, if any, must have been kept stable for at least one month prior to randomization.

Exclusion Criteria:

* History of sensitivity to quetiapine
* Use of antipsychotics, antidepressants, or benzodiazepines (except for short-term use during study as specified in Concomitant Medications section) within one week prior to randomization and throughout the study period.
* Medical conditions that may prevent safe administration of quetiapine including clinically significant hepatic, cardiac, or pulmonary disease.
* Medical disorders that may cause or exacerbate anxiety symptoms.
* Alcohol or drug abuse or dependence within one month of study entry as defined by DSM-IV criteria.
* Schizophrenia, schizoaffective disorder, or bipolar disorder.
* Suicidal or homicidal ideation or other clinically significant dangerousness
* Currently seeking compensation or increase in compensation for the effects of the trauma.
* Initiation or change in psychotherapy within 3 months of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-08; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Global scores on Clinician Administered PTSD Scale - One Week Symptom Version (CAPS-SX) at week 12

SECONDARY OUTCOMES:
Week 12 scores on Positive and Negative Syndrome Scale (PANSS)
Hamilton Depression Rating Scale (HAMD)
Hamilton Rating Scale of Anxiety (HAMA)
Clinical Global Impression Severity Scale (CGI-S)
Clinical Global Impression Improvement Scale (CGI-I)
Davidson Trauma Scale (DTS)
Pittsburgh Sleep Quality Inventory/Pittsburgh Sleep Quality Inventory Addendum (PSQI/PSQI-A)
Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ)
SDS
Arizona Sexual Experience Scale (ASEX)
AIMS
BAS
SAS

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Hamner, MD, Principal Investigator — Ralph H. Johnson VAMC/Medical University of South Carolina
Locations (2):
- United States (2):
  - NM VA Healthcare System, Albuquerque, New Mexico
  - Ralph H. Johnson VAMC, Charleston, South Carolina